CLINICAL TRIAL: NCT02258334
Title: Safety and Immunogenicity Among Adults of Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose, Influenza Vaccines, 2014-2015 Formulations
Brief Title: Study of Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose, Influenza Vaccines in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC55; U1111-1143-8931 (Other: WHO)
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® Quadrivalent, Influenza Vaccine; Fluzone® Intradermal, Influenza Vaccine; Fluzone® High-Dose, Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluzone® Quadrivalent vaccine Group 1 (Experimental): Adults 18 to < 65 years of age randomly assigned to receive an intramuscular injection of Fluzone® Quadrivalent vaccine
  Interventions: Biological: Fluzone® Quadrivalent vaccine, 2014-2015 formulation
- Fluzone® Intradermal vaccine Group 2 (Experimental): Adults 18 to < 65 years of age randomly assigned to receive an intradermal injection of Fluzone® Intradermal vaccine
  Interventions: Biological: Fluzone I®ntradermal vaccine, 2014-2015 formulation
- Fluzone® Quadrivalent vaccine Group 3 (Experimental): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of Fluzone® Quadrivalent vaccine
  Interventions: Biological: Fluzone® Quadrivalent vaccine, 2014-2015 formulation
- Fluzone® High-Dose vaccine Group 4 (Experimental): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of Fluzone® High-Dose vaccine
  Interventions: Biological: Fluzone High Dose vaccine, 2014-2015 formulation

INTERVENTIONS:
Biological: Fluzone® Quadrivalent vaccine, 2014-2015 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent vaccine
  Arms: Fluzone® Quadrivalent vaccine Group 1
Biological: Fluzone I®ntradermal vaccine, 2014-2015 formulation — 0.1 mL, Intradermal
  Other Names: Fluzone® Intradermal vaccine
  Arms: Fluzone® Intradermal vaccine Group 2
Biological: Fluzone® Quadrivalent vaccine, 2014-2015 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent vaccine
  Arms: Fluzone® Quadrivalent vaccine Group 3
Biological: Fluzone High Dose vaccine, 2014-2015 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® High Dose, vaccine
  Arms: Fluzone® High-Dose vaccine Group 4

SUMMARY:
The aim of this trial is to evaluate the safety and immunogenicity of the 2014-2015 formulations of Fluzone® Quadrivalent and Fluzone® Intradermal vaccines in adults 18 to < 65 years or age, and of the 2014-2015 formulations of Fluzone® Quadrivalent and Fluzone® High-Dose vaccines in adults ≥ 65 years of age.

Objectives:

* To describe the safety of the 2014-2015 formulations of Fluzone Quadrivalent and Fluzone Intradermal vaccines in adults 18 to < 65 years of age and the safety of the 2014-2015 formulations of Fluzone® Quadrivalent and Fluzone® High-Dose vaccines in adults ≥ 65 years of age.

Observational objectives:

* To describe the immunogenicity of the 2014-2015 formulations of Fluzone® Quadrivalent and Fluzone® Intradermal vaccines in adults 18 to < 65 years of age and the immunogenicity of the 2014-2015 formulations of Fluzone® Quadrivalent and Fluzone ®High-Dose vaccines in adults ≥ 65 years of age.
* To evaluate the compliance, in terms of immunogenicity, of each study vaccine (Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose) in the applicable age group with the historical requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96.

DETAILED DESCRIPTION:
Adults 18 to < 65 years of age will be randomly assigned in a 1:1 ratio to receive either Fluzone® Quadrivalent or Fluzone® Intradermal vaccine. Adults ≥ 65 years of age will also be randomly assigned in a 1:1 ratio to receive either Fluzone® Quadrivalent or Fluzone® High-Dose vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age on the day of inclusion.
* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* History of serious adverse reaction to any influenza vaccine.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study.
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Prior vaccination with any 2014-2015 formulation of influenza vaccine.
* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone Quadrivalent, Fluzone Intradermal, or Fluzone High-Dose vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information).
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination).
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barré syndrome.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C, as reported by the subject.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug addiction that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 100.4°F) on the day of vaccination. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of an Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of an Investigator or employee with direct involvement in the proposed study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- United States (4):
  - Santa Rosa, California
  - Council Bluffs, Iowa
  - Metairie, Louisiana
  - Cincinnati, Ohio

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 01 October 2014 to 07 November 2014 at 4 clinical sites in the United States.
Pre-assignment Details: A total of 208 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated in this study.
Groups:
- Group 1: Adults 18 to < 65 years of age randomly assigned to receive an intramuscular dose of Fluzone Quadrivalent vaccine.
- Group 2: Adults 18 to < 65 years of age randomly assigned to receive an intradermal dose of Fluzone Intradermal vaccine.
- Group 3: Adults ≥65 years of age randomly assigned to receive an intramuscular dose of Fluzone Quadrivalent vaccine.
- Group 4: Adults ≥65 years of age randomly assigned to receive an intramuscular dose of Fluzone High-Dose vaccine.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 50 | 54 | 52 | 52
Completed | 49 | 54 | 52 | 52
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 3: Adults ≥ 65 years of age randomly assigned to receive an intramuscular dose of Fluzone Quadrivalent vaccine.
- Group 4: Adults ≥ 65 years of age randomly assigned to receive an intramuscular dose of Fluzone High-Dose vaccine.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 50 | 54 | 52 | 52 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 54 | 0 | 0 | 104
  >=65 years | 0 | 0 | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 44.8 (14.9) | 48.0 (12.1) | 73.9 (5.0) | 72.2 (5.4) | 59.8 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 32 | 31 | 127
  Male | 19 | 21 | 20 | 21 | 81
Region of Enrollment [Number; unit: Participants]
  United States | 50 | 54 | 52 | 52 | 208

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Injection-site and Solicited Systemic Reactions Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Injection-site reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering. Grade 3 Injection-site reactions: Pain, Significant, prevents daily activity; Erythema, Swelling, Induration, and Ecchymosis, >100 mm. Grade 3 Systemic reactions: Fever, ≥39.0°C or ≥102.1°F; Headache, Malaise, Myalgia, and Shivering, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 54 | 52 | 52
Percentage of participants
  Injection-site Pain | 53.1 | 51.9 | 36.5 | 40.4
  Grade 3 Injection-site Pain | 0.0 | 1.9 | 0 | 0
  Injection-site Erythema | 6.1 | 35.2 | 3.8 | 7.7
  Grade 3 Injection site Erythema | 0.0 | 0 | 0 | 0
  Injection-site Swelling | 4.1 | 22.2 | 5.8 | 5.8
  Grade 3 Injection-site Swelling | 0.0 | 0 | 0 | 0
  Injection-site Induration | 6.1 | 18.5 | 0 | 1.9
  Grade 3 Injection-site Induration | 0.0 | 0 | 0 | 0
  Injection-site Ecchymosis | 2.0 | 5.6 | 0 | 1.9
  Grade 3 Injection-site Ecchymosis | 0.0 | 0 | 0 | 0
  Fever | 0.0 | 0 | 0 | 0
  Grade 3 Fever | 0.0 | 0 | 0 | 0
  Headache | 28.6 | 18.5 | 17.3 | 25.0
  Grade 3 Headache | 0.0 | 0 | 0 | 1.9
  Malaise | 16.3 | 27.8 | 9.6 | 15.4
  Grade 3 Malaise | 0.0 | 1.9 | 0 | 1.9
  Myalgia | 26.5 | 25.9 | 23.1 | 28.8
  Grade 3 Myalgia | 0.0 | 1.9 | 1.9 | 1.9
  Shivering | 4.1 | 9.3 | 1.9 | 1.9
  Grade 3 Shivering | 0.0 | 0 | 0 | 0

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies to the 2014-2015 Formulation of Fluzone® Quadrivalent or Fluzone® Intradermal or Fluzone® High-Dose Vaccine Antigens Before and Following Vaccination With the Respective Vaccine.
Description: Geometric mean titers of antibodies to Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose vaccine antigens were assessed using the hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Geometric mean titers were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 53 | 52 | 52
Titers (1/dilution)
  A/H1N1; Pre-vaccination (N=49,52,52,52) | 153 [90.6 to 260] | 148 [94.3 to 231] | 148 [96.7 to 226] | 171 [124 to 237]
  A/H1N1; Post-vaccination (N=49,53,52,52) | 707 [490 to 1020] | 632 [459 to 870] | 288 [200 to 414] | 386 [294 to 506]
  A/H3N2; Pre-vaccination (N=49,53,52,52) | 139 [90.9 to 212] | 147 [97.6 to 221] | 168 [119 to 237] | 275 [193 to 390]
  A/H3N2; Post-vaccination (N=49,53,52,52) | 613 [439 to 857] | 648 [470 to 894] | 349 [244 to 499] | 680 [490 to 942]
  B (Yamagata); Pre-vaccination (N=49,53,52,52) | 596 [400 to 888] | 471 [324 to 684] | 471 [342 to 649] | 465 [340 to 635]
  B (Yamagata); Post-vaccination (N=49,53,52,52) | 1836 [1376 to 2449] | 1272 [906 to 1785] | 864 [651 to 1146] | 994 [777 to 1270]
  B (Victoria); Pre-vaccination (N=49,0,52,0) | 252 [164 to 385] | NA [NA to NA] — B (Victoria) antigen was not in the administered vaccine | 273 [195 to 382] | NA [NA to NA] — B (Victoria) antigen was not in the administered vaccine
  B (Victoria); Post-vaccination (N=49,0,52,0) | 1119 [838 to 1495] | NA [NA to NA] — B (Victoria) antigen was not in the administered vaccine | 568 [430 to 750] | NA [NA to NA] — B (Victoria) antigen was not in the administered vaccine

3. Secondary Outcome: Percentage of Participants With Seroprotection Before and Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent or Fluzone® Intradermal or Fluzone® High-Dose Vaccine.
Description: Antibodies to Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose vaccine antigens were assessed using the hemagglutination inhibition (HAI) assay. Seroprotection was defined as a titer ≥40 (l/dilution [dil]) at pre-vaccination and 21 days after vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Seroprotection was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Groups:
- Group 2: Adults 18 to < 65 years of age randomly assigned to receive an intradermal of Fluzone Intradermal vaccine.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 53 | 52 | 52
Percentage of participants
  A/H1N1; Pre-vaccination (N=49,52,52,52) | 77.6 | 84.6 | 82.7 | 90.4
  A/H1N1; Post-vaccination (N=49,53,52,52) | 98.0 | 100.0 | 92.3 | 100.0
  A/H3N2; Pre-vaccination (N=49,53,52,52) | 81.6 | 83.0 | 90.4 | 96.2
  A/H3N2; Post-vaccination (N=49,53,52,52) | 98.0 | 100.0 | 94.2 | 100.0
  B (Yamagata); Pre-vaccination (N=49,53,52,52) | 98.0 | 98.1 | 96.2 | 100.0
  B (Yamagata); Post-vaccination (N=49,53,52,52) | 100.0 | 100.0 | 100.0 | 100.0
  B (Victoria); Pre-vaccination (n=49,0,52,0) | 91.8 | NA — B (Victoria) antigen was not in the administered vaccine | 94.2 | NA — B (Victoria) antigen was not in the administered vaccine
  B (Victoria); Post-vaccination (N=49,0,52,0) | 100.0 | NA — B (Victoria) antigen was not in the administered vaccine | 100.0 | NA — B (Victoria) antigen was not in the administered vaccine

4. Secondary Outcome: Percentage of Participants With Seroconversion Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Antibodies to Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose vaccine antigens were assessed using the hemagglutination inhibition (HAI) assay. Seroconversion was defined as either a pre-vaccination titer < 10 (1/dil) and a post-vaccination titer ≥ 40 (1/dil) or a pre-vaccination titer ≥ 10 (1/dil) and a ≥ 4-fold increase in post-vaccination titer 21 days after vaccination.
Time Frame: Day 21 post-vaccination
Population: Seroconversion was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Groups:
- Group 4: Adults ≥65 years of age randomly assigned to receive an intramuscular dose of Fluzone High Dose vaccine.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 53 | 52 | 52
Percentage of participants
  A/H1N1 (N=49,52,52,52) | 34.7 | 42.3 | 15.4 | 28.8
  A/H3N2 (N=49,53,52,52) | 38.8 | 39.6 | 23.1 | 26.9
  B (Yamagata) (N=49,53,52,52) | 28.6 | 28.3 | 15.4 | 21.2
  B (Victoria) (N=49,0,52,0) | 51.0 | NA — B (Victoria) antigen was not in the administered vaccine | 23.1 | NA — B (Victoria) antigen was not in the administered vaccine

5. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of Antibodies to the 2014-2015 Formulation of Fluzone® Quadrivalent or Fluzone® Intradermal or Fluzone® High-Dose Vaccine Antigens Following Vaccination With the Respective Vaccine
Description: Geometric mean titer ratios of antibodies to Fluzone® Quadrivalent, Fluzone® Intradermal, and Fluzone® High-Dose vaccine antigens were assessed using the hemagglutination inhibition (HAI) assay.
Time Frame: Day 21 post-vaccination
Population: Geometric mean titer ratios were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratios
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 53 | 52 | 52
Titer ratios
  A/H1N1 (N=49,52,52,52) | 4.32 [2.66 to 7.04] | 3.92 [2.54 to 6.06] | 1.91 [1.53 to 2.38] | 2.25 [1.79 to 2.83]
  A/H3N2 (N=49,53,52,52) | 4.26 [2.83 to 6.42] | 4.24 [2.93 to 6.14] | 2.08 [1.65 to 2.62] | 2.48 [1.97 to 3.12]
  B (Yamagata) (N=49,53,52,52) | 3.08 [2.21 to 4.29] | 2.70 [1.95 to 3.74] | 1.83 [1.48 to 2.28] | 2.14 [1.72 to 2.65]
  B (Victoria) (N=49,0,52,0) | 4.39 [3.05 to 6.30] | NA [NA to NA] — B (Victoria) antigen was not in the administered vaccine | 2.08 [1.62 to 2.68] | NA [NA to NA] — B (Victoria) antigen was not in the administered vaccine

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 21 post-vaccination.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/54 | 1/52 | 0/52
Other Adverse Events (participants affected / at risk) | 26/49 | 28/54 | 19/52 | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=49) | Group 2 (N=54) | Group 3 (N=52) | Group 4 (N=52)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=49) | Group 2 (N=54) | Group 3 (N=52) | Group 4 (N=52)
Injection site Pain (General disorders) | 26 (26) | 28 (28) | 19 (19) | 21 (21)
Injection site Erythema (General disorders) | 3 (3) | 19 (19) | 2 (2) | 4 (4)
Injection site Swelling (General disorders) | 2 (2) | 12 (12) | 3 (3) | 3 (3)
Injection site Induration (General disorders) | 3 (3) | 10 (10) | 0 (0) | 1 (1)
Injection site Ecchymosis (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (14) | 10 (10) | 9 (9) | 13 (13)
Malaise (General disorders) | 8 (8) | 15 (15) | 5 (5) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 14 (14) | 12 (12) | 15 (15)
Shivering (General disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications